CLINICAL TRIAL: NCT01416727
Title: A Randomised Trial of Simulation Training vs Workplace-Based Supervision for Junior Doctors in Psychiatry
Brief Title: Simulation Training vs Workplace-Based Supervision in Psychiatry
Acronym: EPIC-OSkER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); South London and Maudsley Charitable Funds (Unknown); South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Dr Amy C Iversen, King's College London
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2011/051
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-08

CONDITIONS: Clinical Skills Training
Keywords: Patient Simulation; Education, Medical, Graduate; Internship and Residency; Psychiatry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSkER (Experimental): "Observed SKills in the Emergency Room" - workplace-based supervision.
  Interventions: Other: Observed SKills in the Emergency Room
- EPIC (Experimental): "Emergency Psychiatry Immersion Course" - simulation-based training.
  Interventions: Other: Emergency Psychiatry Immersion Course

INTERVENTIONS:
Other: Emergency Psychiatry Immersion Course — A two-day simulation-based training course covering assessment of self-harm, capacity, managing aggression, working with the emergency team and medical emergencies in the psychiatric hospital
  Arms: EPIC
Other: Observed SKills in the Emergency Room — For four weeks, participants will be accompanied by a senior psychiatric registrar or consultant psychiatrist, who has received training in giving feedback, during their on-call duties. Each participant will receive between 8-12 hours of 1:1 training.
  Arms: OSkER

SUMMARY:
The purpose of this study is to evaluate and compare the effectiveness of two forms of clinical skills training for teaching emergency psychiatry skills to doctors who have just started to work in psychiatry

DETAILED DESCRIPTION:
Junior doctors starting work in psychiatry soon encounter a number of situations in the workplace for which they have had little or no preparation either at medical school or from work in other specialities. They will encounter clinically complex situations such as rapid tranquillisation, crisis presentations of self-harm, suicide risk assessment, overseeing supervised confinement and making decisions to admit or discharge mentally ill patients. Furthermore, many of these situations occur out of hours when there is little direct senior supervision available. The traditional induction programme is delivered in a didactic format, which does not encourage effective learning, nor does it allow any opportunity to practise or acquire hands-on skills or non-technical skills such as interprofessional communication, leadership and situational awareness. In the interests of patient safety and improving the quality of care and patient's experience, there is an urgent need to identify ways of improving induction and quickly equipping junior doctors with the clinical skills necessary to practise safely in psychiatry. We propose to evaluate and compare two approached to improved skills training in psychiatry: 1. workplace-based observation and feedback; 2. simulation training.

All new junior doctors starting work in the South London and Maudsley NHS Foundation Trust, London, UK, in August 2011 will be invited to take part in a randomised controlled trial of training in addition to the standard induction. Following a day of lectures on relevant clinical topics, participants will be randomly allocated to receive either observed workplace-based training by a more senior doctor during their on-call duties, or a two-day simulation-based training course. Before and after the training, assessments of participants' clinical skills and attitudes will be carried out by questionnaires and by observations of simulated clinical encounters. Changes in performance will be compared between the two groups. Longer term evaluation will be carried out by means of qualitative interviews and simulated clinical encounters once participants have been working for several months.

ELIGIBILITY:
Inclusion Criteria:

* Junior doctors starting work at the South London and Maudsley NHS Foundation Trust in August 2011 in any of the following grades: 1. Core Psychiatric Training; 2. Foundation Training; 3. General Practice Vocational Training; 4. Core Trainee 1-3 equivalent posts, e.g. long-term locums

Exclusion Criteria:

* Unwillingness to participate in the study
* Inability to attend the training programme or participate in the evaluation

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Change in global clinical skills | Baseline; 4 weeks; 16 weeks
  Participants will participate in a single simulated clinical encounter. Encounters will be video-recorded and then rated by observers, who are blind to the allocation status and time point of each video, using a global rating scale.

SECONDARY OUTCOMES:
Change in technical clinical skills | Baseline; 4 weeks; 16 weeks
  Participants will participate in a single simulated clinical encounter. Encounters will be video-recorded and then rated by observers, who are blind to the allocation status and time point of each video, using a checklist-based rating scale.
Change in attitudes towards teamworking | Baseline; 4 weeks; 16 weeks
  The Operating Room Management Attitudes Questionnaire will be modified to be appropriate for working in psychiatry.
Change in attitudes towards self-harm | Baseline; 4 weeks; 16 weeks
  The Attitudes to Deliberate Self-Harm Questionnaire
Self-reported views on usefulness and acceptability of the training programmes | 4 weeks
  Post-course feedback questionnaire
Qualitative evaluation | 8 - 12 weeks
  Focus groups will be conducted to evaluate how participants have learned to manage psychiatric emergencies, and the contribution of the courses to their learning.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry, King's College London, London, United Kingdom